CLINICAL TRIAL: NCT02005146
Title: Retrospective Observational Study to Define HBsAg Loss With or Without Seroconversion to antiHBs in Patients With Chronic Hepatitis by B Virus Treated With Nucleoside/Nucleotide Analogs
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: ESG-HEP-2013-01
Record Dates: First submitted 2013-11-15; First posted 2013-12-09 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis B Treated With Nucleoside/Nucleotide Analogues
Keywords: Hepatitis B; Nucleoside/nucleotide; HBsAg loss
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis B treated with nRTI: Patients with chronic hepatitis B with HBsAg loss treated with nucleoside/nucleotide analogues (Lamivudine, Adefovir, Tenofovir, Telbivudine, Entecavir, Emtricitabine)

SUMMARY:
Define the patients who lost HBsAg, studying the loss predictive factors and if there was suspension of treatment, study the evolution after that

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Chronic hepatitis B (HBeAg+ or HBeAg-)
* HBsAg loss
* Treated with nucleoside/nucleotide analogues
* With or without previous interferon (IFN/PEG-IFN)
* Patients with HBsAg loss after 2006
* Immunocompetent patients

Exclusion Criteria:

* Spontaneous HBsAg loss
* HBsAg loss while treatment in monotherapy or combinated with IFN or PEG-IFN.
* Patients with hepatitis delta virus (HDV) coinfection.
* Patients with hepatitis C virus (HCV) coinfection.
* Patients with HIV coinfection.
* Patients with liver transplant.
* Patients with reactivated hepatitis B virus (HBV) by immuno-suppressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B with HBsAg loss treated with nucleoside/nucleotide analogues
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Epidemiological characteristics from hepatitis B patients who lost HBsAg related to treatment with nucleoside/nucleotide analogues | 15 months
  Study the number of diferents virological, serological, clinical, histological, biochemical characteristics from hepatitis B patients who lost HBsAg related to treatment with nucleoside/nucleotide analogues.

SECONDARY OUTCOMES:
Epidemiological characteristics in case of suspension of treatment. | 15 months
  Count the diferents characteristics virological, histological, serological, and the clinical course of this patients whom must to be suspended the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Suárez García, Principal Investigator — Hospital Universitario Virgen de Valme; Miguel Ángel Simón Marco, Principal Investigator — Hospital Clínico Universitario Lozano Blesa
Locations (22):
- Spain (22):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario Santiago, Santiago de Compostela, La Coruña
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Torrecárdenas, Almería
  - Hospital Clínic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital de Navarra, Pamplona
  - Hospital Donosti, San Sebastián
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital General Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza